CLINICAL TRIAL: NCT05584189
Title: Over the Counter Rapid Antigen Test for Detection of SARS-CoV-2 Virus: Human Usability Study
Brief Title: COVID-19 MP Biomedicals Rapid SARS-CoV-2 Antigen Test Usability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MP Biomedicals, LLC (Industry)
Collaborators: New Day Diagnostics (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDP-SOP-TNC-013
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-10

CONDITIONS: Sars-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open-label, prospective study to evaluate the usability of the Rapid SARS-CoV-2 Antigen Test when a lay person conducts the test on themselves or another study participant. Potential subjects will be those presenting for COVID-19 testing. The study will evaluate the layperson usability of the Rapid SARS-CoV-2 Antigen Test by assessing the performance of the Rapid SARS-CoV-2 Antigen Test under the supervision of qualified site personnel, as well as having the testing participant complete assessments measuring .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- At least 30 persons 14-65+ years of age who test themselves (Experimental): Participants between the ages of 14-65+ years will perform candidate Ag self-test kit anterior nasal specimen collection and testing under the supervision of qualified site personnel in person.
  Interventions: Device: Rapid SARS-CoV-2 Antigen Test
- At least 30 persons 18-65+ years of age who test another participant (Experimental): Participants between the ages of 18-65+ years will perform candidate Ag self-test kit anterior nasal specimen collection on another participant aged 2-65+ years and testing of the candidate Ag self-test kit under the supervision of qualified site personnel in person.
  Interventions: Device: Rapid SARS-CoV-2 Antigen Test

INTERVENTIONS:
Device: Rapid SARS-CoV-2 Antigen Test — Candidate Ag self-test kit anterior nasal specimen collection and testing will be done under the supervision of qualified site personnel in person.

SUMMARY:
SARS-CoV-2 rapid antigen over the counter usability study.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is a disease caused by a newly discovered coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The SARS-CoV-2 is a β-coronavirus, which is enveloped non-segmented positive-sense RNA virus 2. It is spread by human-to-human transmission via droplets or direct contact, and infection has been estimated to have mean incubation period of 6.4 days and a basic reproduction number of 2.24-3.58. Among patients with pneumonia caused by SARS-CoV-2, fever was the most common symptom, followed by cough. On 11 March 2020, the COVID-19 outbreak was characterized as a pandemic by the WHO. Since then, over 70 million people worldwide have been infected with the virus with over 1.5 million deaths attributed to the virus5. Laboratory testing for SARS-CoV-2 is currently being performed to determine if an individual has active infection via detection of viral RNA or if an individual has an immune response to the virus from a previous infection via detection of antibodies.

Specimen collection is a crucial first step in the evaluation of an individual's SARS-CoV-2 infection status. The goal of this project is to evaluate human usability of a rapid SARS-CoV-2 antigen test for over the counter (OTC) use. Study subjects under EDP supervision, either in-person or via video conference, will collect and test anterior nasal swab samples. The Rapid SARS-CoV-2 Antigen Test collection and testing methodology is viewed as a convenient and inexpensive method to test clinical specimens for SARS-CoV-2 and OTC access will improve the availability of COVD-19 testing.

The COVID-19 Antigen Rapid Test Device detects SARS-CoV-2 viral antigens through visual interpretation of color development. Anti-SARS-CoV-2 antibodies are immobilized on the test region of the nitrocellulose membrane. Anti-SARS-CoV-2 antibodies conjugated to colored particles are immobilized on the conjugated pad. A sample is added to the extraction buffer which is optimized to release the SARS-CoV-2 antigens from specimen. During testing, the extracted antigens bind to anti-SARS-CoV-2 antibodies conjugated to colored particles. As the specimen migrates along the strip by capillary action and interacts with reagents on the membrane, the complex will be captured by the anti-SARS-CoV-2 antibodies at the test region. Excess colored particles are captured at the internal control zone. The presence of a colored band in the test region indicates a positive result for the SARS-CoV-2 viral antigens, while its absence indicates a negative result. A colored band at the control region serves as a procedural control, indicating that the proper volume of specimen has been added and membrane wicking is working. (See Appendix 1).

ELIGIBILITY:
Inclusion Criteria:

* The study population will include subjects from 2 years old to greater than 65 years old.
* Lay subjects who perform the test on themselves must be able to read, write, speak, and understand English or Spanish.

Exclusion Criteria:

* Participants who regularly use home diagnostic tests, such as glucose meters, will be excluded.
* Persons under 2 years of age will be excluded from participation.
* Persons under 14 years of age will be excluded from performing the Rapid SARS-CoV-2 Antigen Test on themselves.
* Persons under 18 years of age will be excluded from performing the Rapid SARS-CoV-2 Antigen Test on another qualified participant.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Liggett, PhD, Principal Investigator — New Day Diagnostics
Locations (1):
- EDP Biotech Corporation, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- See also: Johns Hopkins University Center for Health Security Website. 2020. — https://www.centerforhealthsecurity.org
- See also: WHO. 2022 — https://www.who.int/

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Who Test Themselves: Participants between the ages of 14-65+ years will perform candidate Ag self-test kit anterior nasal specimen collection and testing under the supervision of qualified site personnel in person.
  Rapid SARS-CoV-2 Antigen Test: Candidate Ag self-test kit anterior nasal specimen collection and testing will be done under the supervision of qualified site personnel in person.
- Participants Who Test Another Participant: Participants between the ages of 18-65+ years will perform candidate Ag self-test kit anterior nasal specimen collection on another participant aged 2-65+ years and testing of the candidate Ag self-test kit under the supervision of qualified site personnel in person.
  Rapid SARS-CoV-2 Antigen Test: Candidate Ag self-test kit anterior nasal specimen collection and testing will be done under the supervision of qualified site personnel in person.
Period: Overall Study
Arm/Group | Participants Who Test Themselves | Participants Who Test Another Participant
Started | 53 | 46
Completed | 53 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | At Least 30 Persons 14-65+ Years of Age Who Test Themselves | At Least 30 Persons 18-65+ Years of Age Who Test Another Participant | Total
Number analyzed (Participants) | 53 | 46 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 0 | 6
  Between 18 and 65 years | 45 | 42 | 87
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 27 | 22 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 49 | 42 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 5 | 17
  White | 37 | 34 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: 30 Candidate Ag Test Self-collections
Description: Lay subjects aged 14-65+ who will perform collection of the candidate Ag self-test kit on themselves under the supervision of qualified site personnel in person.
Time Frame: One Hour
Population: The second arm of the trial was analyzed under the second primary outcome measure. This is why the number is 0 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | At Least 30 Persons 14-65+ Years of Age Who Test Themselves | At Least 30 Persons 18-65+ Years of Age Who Test Another Participant
Number analyzed (Participants) | 53 | 0
Participants | 53 | 0

2. Primary Outcome: 30 Candidate Ag Test Collections of Another
Description: Lay subjects aged 18-65+ who will perform collection of the candidate Ag self-test kit on another participant aged 2-65+ years under the supervision of qualified site personnel in person
Time Frame: One Hour
Population: The first arm of the trial was analyzed under the first primary outcome measure. This is why the number is 0 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | At Least 30 Persons 14-65+ Years of Age Who Test Themselves | At Least 30 Persons 18-65+ Years of Age Who Test Another Participant
Number analyzed (Participants) | 0 | 46
Participants | 0 | 46

3. Secondary Outcome: At Least One Enrollment of a Spanish Speaking Lay User
Description: At least one lay subject aged 14-65+ who will perform collection of the candidate Ag self-test kit on themselves under the supervision of qualified site personnel in person and/or at least one lay subject aged 18-65+ who will perform collection of the candidate Ag self-test kit on another participant aged 2-65+ years under the supervision of qualified site personnel in person.
Time Frame: One Hour
Measure: Count of Participants; unit: Participants
Arm/Group | At Least 30 Persons 14-65+ Years of Age Who Test Themselves | At Least 30 Persons 18-65+ Years of Age Who Test Another Participant
Number analyzed (Participants) | 53 | 46
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: One hour
Arm/Group | At Least 30 Persons 14-65+ Years of Age Who Test Themselves | At Least 30 Persons 18-65+ Years of Age Who Test Another Participant
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/46
Other Adverse Events (participants affected / at risk) | 0/53 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT05584189/Prot_000.pdf
  • Informed Consent Form: Minor Assent Form (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05584189/ICF_001.pdf
  • Informed Consent Form: Adult Consent Form (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05584189/ICF_003.pdf